CLINICAL TRIAL: NCT01758965
Title: Surgicel® (Fibrillar) for Preventing Delayed Bleeding After ESD in Stomach: A Prospective Randomized Study
Brief Title: Surgicel® Fibrillar for Delayed Bleeding After ESD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Su Jin Hong, MD, PhD, Soonchunhyang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MD_SCHBC_IRB_2012-06
Record Dates: First submitted 2012-12-27; First posted 2013-01-01 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Benign Neoplasm of Stomach; Malignant Neoplasm of Stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — Surgicel

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- combination therapy of H2RA and surgicel (Experimental): H2RA and surgicel
  Interventions: Other: H2RA and surgicel
- Monotherapy of PPI (Experimental): PPI
  Interventions: Other: PPI

INTERVENTIONS:
Other: PPI — monotherapy of PPI
  Arms: Monotherapy of PPI
Other: H2RA and surgicel — combination therapy of H2RA and surgicel
  Arms: combination therapy of H2RA and surgicel

SUMMARY:
The aim of this study is to assess the effect of Surgicel® Fibrillar as adjuvant treatment to H2RA on preventing ulcer bleeding after ESD for gastric epithelial tumors

DETAILED DESCRIPTION:
1. Patient (1) Inclusion: Diagnosed as gastric dysplasia or early gastric cancer

   * Scheduled for ESD (2) Exclusion: Coagulopathy- liver cirrhosis, thrombocytopenia
   * Anti-platelet agents
2. Method

(1) Study group: combination with Surgicel® Fibrillar and H2RA (2) Control group: monotherapy with PPI 3. Sample size : 157 4. Result

1. Primary endpoint: rate of delayed bleeding after ESD
2. Secondary endpoint: follow-up hemoglobin after ESD

ELIGIBILITY:
Inclusion Criteria:

* ESD for gastric dysplasia or early gastric cancer

Exclusion Criteria:

* Coagulopathy: liver cirrhosis, thrombocytopenia
* Anti-platelet agents

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Delayed bleeding rate after ESD | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Digestive Disease Center, Department of Internal Medicine, Soonchunhyang University College of Medicine, Bucheon-si, Gyeonggi-do, South Korea